CLINICAL TRIAL: NCT06459778
Title: A Single-center Randomized Controlled Trial on Piezo-ICSI Improving Oocyte Fertilization and Embryo Development in Elderly Infertile Patients
Brief Title: Piezo-ICSI to Improve the Developmental Potential of Fertilized Oocytes in Aged Infertility Women With Assisted Reproductive Technology
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Wang Shanshan, Reseaerch fellow, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SZ-Piezo-1
Record Dates: First submitted 2024-06-03; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Infertility, Female; Intracytoplasmic Sperm Injections
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Piezo-ICSI group, Oocytes in this group will be fertilized with Piezo-ICSI (Experimental): The Piezo-ICSI technique involves the use a piezoelectric actuator to create high speed movement of the injection pipette. These fine movements allow precise microdrilling of the zona and smooth penetration of injection pipette into the cytoplasm and a single Piezo pulse facilitates breakage of the membrane, with the spermatozoa deposited into the cytoplasm without the need for cytoplasmic aspiration or agitation. Since the initial reports of the use of Piezo-ICSI in human oocytes, there have been notable improvements made to the technique, including a change in the operating fluid, leading to a safe and effective technique suitable for clinical use. In addition, when this technology was utilized in patients with poor outcomes, including low fertilization, high degeneration or low utilization in previous cycles, it resulted in improved fertilization, degeneration, embryo utilization and pregnancy rates compared with conventional ICSI.
  Interventions: Device: Piezo-ICSI
- Control group, Oocytes in this group will be fertilized with conventional ICSI (No Intervention)

INTERVENTIONS:
Device: Piezo-ICSI — Participants had their oocytes cohort divided, where half were injected using conventional ICSI and the other half were injected using Piezo-ICSI.
  Arms: Piezo-ICSI group, Oocytes in this group will be fertilized with Piezo-ICSI

SUMMARY:
The goal of this clinical trial is to test Piezo-ICSI on improving oocyte fertilization and embryo development in elderly infertile patients undergoing intracytoplasmic sperm injection (ICSI). The main question it aims to answer is whether Piezo-ICSI could improve oocyte fertilization and embryo development. Participants requested ICSI are asked to randomly culture equal numbers of oocyte and embryo with or without Piezo-ICSI. At the time of injection, two or more mature oocytes were split into two groups (i) conventional ICSI and (ii) Piezo-ICSI (50:50 split).

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all participants will write the informed contents. This study is a randomized controlled study compare different ICSI methods on the fertilization and embryo development. Sibling oocytes were randomly divided into test group (Piezo-ICSI) and control group (conventional ICSI).

Specific method of randomization: all the oocytes of each subject were distributed into two dishes (dish 1 and dish 2). If the oocyte number is odd, put the extra oocyte into dish 1. Using statistical software, the two dishes were randomly treated as test group and control group. Thus, a random allocation table was generated and a separate random envelope was made for each subject. The random envelope is kept and distributed by the relevant personnel who are not involved in the screening and treatment of subjects and are authorized by the researcher. Each selected subject must open the random envelope. The subjects were subjected to routine ovulation promotion, and then the acquired oocytes and cumulus cell complexes (COCs) were obtained and fertilized in vitro. The test group oocytes were fertilized with Piezo-ICSI, while the control oocytes were fertilized with conventional ICSI.

Thus, half of the oocytes from each elderly infertile patient were treated with Piezo-ICSI.

ELIGIBILITY:
Inclusion Criteria:

1. 35 years ≤ age ≤ 42 years;
2. Number of IVF/ICSI cycles ≤ 2

Exclusion Criteria:

1. Egg donor cycle
2. Chromosome abnormality;
3. Adenomyosis, hysteromyoma, thin endometrium, endometriosis and other uterine diseases;
4. Patients with repeated implantation failure

Ages: 35 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 147 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
fertilization rate post intracytoplasmic sperm injection | 16-18 hours post intracytoplasmic sperm injection
  The primary outcome measure was the fertilization rate 16-18 hours post intracytoplasmic sperm injection

CONTACTS AND LOCATIONS:
Locations (1):
- Reproductive Medicine Center, The affiliated Drum Towel Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No